CLINICAL TRIAL: NCT06142448
Title: Unravelling the Neural Mechanisms Underlying Compensation Strategies for Gait Impairments in Parkinson's Disease: a Transnational, Multimodal Approach
Brief Title: The Effect of Compensation Strategies on Gait Impairment in Parkinson's Disease
Acronym: UNITE-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: KU Leuven (Other); Tel-Aviv Sourasky Medical Center (Other Government); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 113692
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Rehabilitation; Gait Impairment; Personalized treatment; Compensation strategies
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Responders (Experimental)
  Interventions: Device: Cueing app
- Non-responders (No Intervention)

INTERVENTIONS:
Device: Cueing app — All participants that are included come to the movement lab for the baseline measurement. The baseline measurement consists out of extensive clinimetrics (for example MDS-UPDRS) to identify patient characteristics. With the use of an objective gait assessment, the effectiveness of both internal and external cueing is determined. This will divide the participants in three groups; responders, non-responders and in between. Participants who clearly respond to either internal or external cueing (determined as the responders) are asked to apply the working form of cueing in daily life during the six-month follow-up. During this period the participants will use a mobile application that can provide them with a rhythmic auditory stimulus and records the use of this application.
  After 6 months, both the responders and non-responders are asked to return to the lab for the follow up measurement in which the baseline measurement is repeated to evaluate the effect of long-term cueing.
  Arms: Responders

SUMMARY:
Gait disturbances are disabling and common in Parkinson's disease (PD). Patients use many different, and typically self-developed, strategies to compensate for their walking abnormalities. There is a wide variety of compensatory strategies, of which external and internal cueing are the most commonly known. External cueing refers to externally produced predictive stimuli such as a metronome, whereas internal cueing refers to a movement reference generated internally, such as counting while walking. The efficacy of external and internal cueing varies dramatically across patients, and some patients can even be identified as 'non-responders' to a particular cue. Consequently, a one-size-fits-all approach simply does not suffice, which increases the need for better understanding of the key mechanisms behind these compensation strategies. Furthermore, it is still unknown how the efficacy of compensation strategies changes longitudinally. The goal of the UNITE-PD project is to address these questions. The investigators aim to investigate whether the efficacy of internal and external cueing changes over time, and whether it is differentially affected in responders and non-responders. In order to work towards a more personalized treatment for patients with PD, the investigators also aim to identify potential patient characteristics that can mediate the actual use of compensation strategies in daily life.

The multicenter UNITE-PD project is divided in a joint package and individual site-specific packages. All partners will investigate the neural working mechanisms of compensation strategies in PD from different angles in the site-specific packages. The joint package focusses on the long-term effect of the compensation strategies and the potential patient characteristics that can influence the efficacy of the compensation strategies. In this project, the investigators will define responders and non-responders to external and/or internal cueing. With the use of extensive clinimetrics, the aim is to identify patient characteristics that might influence the efficacy. With the use of a custom made cueing app (which will be applied during a follow up period of six months), the long-term effect of cueing in the responders can be investigated.

Together, all centers aim to include a total of 384 participants (Netherlands N = 104, Belgium N =90, Israel N = 75, Italy N = 115). Importantly, this sample size is not based on the joint workpackage described here, but on the numbers needed for the individual site-specific work packages.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of age > 18 years with idiopathic Parkinson's disease;
* Written informed consent.

Exclusion Criteria:

* Daily usage of compensation strategies for the past month;
* Presence of deep brain stimulation (DBS);
* Presence of severe co-morbidity limiting ambulation (e.g. stroke, orthopaedic problems);
* Inability to walk unaided (with the exception of a customary cane);
* Inability to walk for > 3 minutes consecutively;
* Severe auditory impairments, hampering perception of auditory cues;
* Severe cognitive impairment (MMSE < 21)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Gait Variability | Six months
  Gait variability defined as the coefficient of variation of stride time. We will compare gait variability between the baseline condition, and the cueing conditions.

SECONDARY OUTCOMES:
Gait speed | Six months
  Gait speed defined in meters per second

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands